CLINICAL TRIAL: NCT05604339
Title: Etude de la récupération et Des Modifications de la rhéologie Sanguine Chez Les Coureurs d'Ultraendurance ERUPTION-3 / Study of Recovery and Blood Rheology Changes in Ultra-endurance Runners ERUPTION-3
Brief Title: Study of Recovery and Blood Rheology Changes in Ultra-endurance Runners (ERUPTION-3)
Acronym: ERUPTION-3
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Jean Monnet University (Other); Aspetar Orthopedic and Sports Medicine Hospital (Unknown); Universite de La Reunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/18
Record Dates: First submitted 2022-10-03; First posted 2022-11-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While the acute consequences of an ultratrail are beginning to be well documented, data on the study of recovery in the aftermath of an event are much rarer.

In order to overcome these various limitations, the main study of the ERUPTION-3 project is set up on the Grand Raid de La Réunion 2022 races.

In the context of exercise responses, the rheological properties of blood can impact the endurance performance. In contrast to short-distance events, the study of blood rheology and red blood cells integrity in long-distance events such as ultra-endurance races is poorly documented in the literature.

In the ancillary study, the work that is intended to be carried y out will complement the initial results found by a previous research on 23 runners during the Ultra Trail du Mont Blanc. This ancillary study will also be an opportunity to complete the data from the main study by studying the kinetics of biomarker recovery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Participating in the Grand Raid de la Réunion race (Mascareignes, Trail de Bourbon or Diagonale des fous)
* Affiliated or beneficiary of a social security scheme
* Not opposed to the research for the main study
* Having given their written consent for the participants of the ancillary study

Exclusion Criteria:

* Not understanding French
* Protected adult (guardianship or curatorship) or under court protection
* Who have difficulty swallowing paracetamol capsules and for whom it will therefore be difficult to swallow the e-Celsius® Performance capsules (for the ancillary study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the main study, the recruitement of 1300 participants within the 6500 runners of the Grand Raid is planned. Call for volonteers will be made via the association organising the race. For the ancillary study, among these 1300 participants, 90 will be choosen (30 of each race, Diagonale des Fous, Trail de Bourbon and Mascareignes) to participate to this optional study.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Recovery and its kinetics in the aftermath of an ultratrail run in a tropical environment. | 3 Months
  Evaluate by means of subjective evaluations in the aftermath of an ultratrail run in a tropical environment:
  - Hooper Index (4 questions: sleep, stress, tiredness and muscular pain) each ranging from 1 to 7 with 1 being very good ranking and 7 worse ranking
Recovery and its kinetics in the musculo-articular evaluations in the aftermath of an ultratrail run in a tropical environment. | 3 Months
  Evaluate by means of subjective evaluations in the aftermath of an ultratrail run in a tropical environment:
  - musculo-articular recovery (descriptive assessment no score)
Recovery and its kinetics of sleep in the aftermath of an ultratrail run in a tropical environment. | 3 Months
  Evaluate by means of subjective evaluations in the aftermath of an ultratrail run in a tropical environment:
  - sleep questionnaire (descriptive assessment no score)
Recovery and its kinetics of tiredness in the aftermath of an ultratrail run in a tropical environment. | 3 Months
  Evaluate by means of subjective evaluations in the aftermath of an ultratrail run in a tropical environment:
  - tiredness questionnaire (descriptive assessment no score)
Recovery and its kinetics of injury in the aftermath of an ultratrail run in a tropical environment. | 6 Months
  Evaluate by means of subjective evaluations in the aftermath of an ultratrail run in a tropical environment:
  - injury questionnaire (descriptive assessment no score)
To evaluate recovery and its kinetics in its different dimensions in ultra-endurance runners | 1 Month
  Evaluate by means of objective evaluations in the aftermath of an ultratrail run in a tropical environment:
  1200m and 400m test (best race time)
Ancillary Study: Change in Hematological Recovery biomarkers | Day 2, Day 5, Day 9 and Day 16
  Evaluate the changes in recovery kinetics of biological markers (hematological:haemoglobin in g/dL ) directly after the race in comparison with measurements taken before the race
Ancillary Study: Change in Muscular Recovery biomarkers | Day 2, Day 5, Day 9 and Day 16
  Evaluate the changes in recovery kinetics of biological markers (muscular: Creatin PhosphoKinase in UI/L), directly after the race in comparison with measurements taken before the race
Ancillary Study: Change in Inflammatory Recovery biomarkers | Day 2, Day 5, Day 9 and Day 16
  Evaluate the changes in recovery kinetics of biological markers (inflammatory: Protein C-reactive in mg/L) directly after the race in comparison with measurements taken before the race
Ancillary Study: Change in Hepatic Recovery biomarkers | Day 2, Day 5, Day 9 and Day 16
  Evaluate the changes in recovery kinetics of biological markers (hepatic: ASAT & ALAT in UI/L) directly after the race in comparison with measurements taken before the race
Ancillary Study: Blood rheologic properties and the senescence of red blood cells | Post-race (between day2 and day4 depending on the time of race arrival)
  Evaluate the rheologic biomarkers by measuring the blood viscosity directly after the race in comparison with measurements taken before the race
Ancillary Study: Senescence of red blood cells | Post-race (between day2 and day4 depending on the time of race arrival)
  Evaluate the Senescence of red blood cells directly after the race in comparison to before the race, by taking blood samples and analysing them using spectrophotometry and fluorescent-activated cells sorting

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOUSCAREN, Principal Investigator — CHU La Réunion
Locations (1):
- CHU de la Réunion, Saint-Denis, Reunion